CLINICAL TRIAL: NCT02709694
Title: Imaging Biomarkers in Crohn's Associated Spondyloarthritis
Acronym: MaRCH-on
Status: Completed | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-491
Record Dates: First submitted 2016-02-24; First posted 2016-03-16 (Estimated); Results first posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-09

CONDITIONS: Crohn's Disease; Spondyloarthritis
MeSH Terms: conditions — Crohn Disease; Spondylarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood for C-reactive Protein and stool samples for fecal microbial 16s rRNA sequencing
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — No drug or device intervention. However, participants will receive MRI of their spine, answer questionnaires, provide clinical history as well as blood and stool sample. Joint exams will also be performed on all participants.

SUMMARY:
In patients with Crohn's Disease, symptoms of inflammatory back pain (IBP) precede changes on plain X-rays by years, and MRI changes of axial inflammation precede development of X-ray changes. Sacroiliitis on MRI without x-ray changes (i.e.Non radiographic SpA) is a valid diagnostic criterion for Spondyloarthritis (SpA) and leads to earlier diagnosis of SpA in patients with IBP. It is unclear when MRI changes occur, and if they precede clinical symptoms of IBP. There are reports of asymptomatic sacroiliitis noted on MRI in Crohn's patients. This is important, as MRI evidence of inflammation may be the first sign of incipient SpA. Inflammation in other regions of the axial skeleton in SpA patients has also been documented, but its significance is unknown. The prospect of undiagnosed and untreated inflammation is concerning, as it can lead to significant morbidity. Moreover, relationship between MRI evidence of axial inflammation-likely a proxy for systemic inflammation- and patient reported outcomes (e.g. ASDAS-CRP= Ankylosing Spondylitis Disease Activity Score- C reactive protein, BASDAI= Bath Ankylosing Spondylitis Disease Activity Index, SF-12 = Short Form- 12, HBI= Hervey Bradshaw Index and PROMIS-29= Patient Reported Outcome Measurement Information System-29), has not been reported. Recent unpublished data from Dr. Longman's lab (collaborator) suggest a distinct intestinal dysbiosis in Crohn's associated SpA. But relationship between this microbiome and MRI changes is yet to be determined.

Identifying inflammation earlier on MRI- in the absence of clinical symptoms will provide an opportunity to intervene early with available therapies, such as- biologics etc. Asymptomatic MRI changes could be a marker of underlying systemic inflammation- which is a risk factor for poor outcomes in Crohn's associated SpA. Studying association between whole spine MRI changes with patient reported outcomes) may facilitate informed clinical decision making to initiate targeted therapy to prevent progression of structural damage. Understanding microbial dysregulation in this population, and correlation with MRI changes, could lead to development of therapy targeted to restore intestinal symbiosis.

DETAILED DESCRIPTION:
IMAGING AND CROHN'S ASSOCIATED SpA: Crohn's disease (CD) is the most common type of inflammatory bowel disease (IBD). It affects an estimated 0.7 million patients in United States and is responsible for 0.2 million hospitalizations each year.1 Although the gastrointestinal tract is the primary site of inflammation, inflammatory arthritis (both peripheral and axial) can affect between 12.8-23% of patients with Crohn's Disease2,3, and axial SpA alone has been reported to effect 6.7% to 18% of Crohn's patients.4 However, in 2 recent studies5,6, radiological sacroiliitis was reported to be present in 27% and 52% in IBD patients. MRI changes of inflammation precede radiological sacroiliitis by years but it is not clear when this occurs. Presence of damage on x-ray in asymptomatic patients may suggest that Crohn's associated axial SpA could be underdiagnosed. Since Crohn's associated SpA often affects younger patients, undertreatment or missed diagnoses could have a significant impact on health related quality of life (HR-QoL) and disability during prime wage earning and child rearing years.7

"Non-radiographic axial spondyloarthritis" is a term used to describe patients with symptomatic SpA who do not have findings on plain x-rays. These patients can have identical symptoms to those with radiographic evidence of cartilage loss and erosions, and anti-TNF (anti-Tumor Necrosis Factor) therapy has been shown to be effective in those with non-radiographic SpA.8 These patients are a clinically relevant subgroup, as 20% of patients with only MRI evidence of sacroiliitis will progress to non-reversible radiographic SpA over two years.9 Therefore, MRI evidence of sacroiliitis, in conjunction with inflammatory back pain is now sufficient to diagnosis SpA. In fact, MRI imaging is a standard component of current SpA diagnostic criteria, (ASAS: Assessment of SpondyloArthritis International Society),10 and MRI changes of sacroiliitis are routinely used to identify SpA patients for clinical trials.11

However, despite these new definitions there is a deficiency of published research evaluating the clinical significance of MRI findings in patients with Crohn's disease. Of all the SpA-associated diseases, Crohn's-associated SpA has a particularly high burden of extra-articular inflammation. Studies suggest only half to two thirds of patients with CT or MRI evidence of inflammation have symptoms of inflammatory back pain.1,12 This suggests that in Crohn's disease, MRI imaging biomarkers may be identifying early disease, analogous to the way that ultrasound can identify subclinical rheumatoid arthritis.13 We therefore hypothesize that in a mixed cohort of Crohn's patients with and without inflammatory back pain, MRI imaging biomarkers will correlate with measures of health status which reflect systemic inflammatory burden, (i.e. BASDAI, SF-12) independent of symptoms of inflammatory back pain.

MRI IMAGING BIOMARKERS: A POTENTIAL CARDIOVASCULAR RISK FACTOR? The observed discordance between axial inflammation seen on MRI and inflammatory back pain raises a particularly intriguing clinical question: could Crohn's patients with imaging evidence of axial inflammation but without axial symptoms potentially benefit from therapy?

It is very well established that in rheumatoid arthritis and psoriatic arthritis, systemic inflammation is associated with myocardial infarction, stroke and death, and that treating inflammation improves cardiovascular outcomes.14,15.

Recent population based study from Europe and Canada showed increased risk of cardiovascular mortality in patients with Ankylosing Spondylitis.16,17 Despite clear evidence that cardiovascular risk is increased in SpA, how to quantify the increased risk is not straightforward. There is no consistently reliable marker of systemic inflammation in these patients; sedimentation rate (ESR) and C-reactive protein (CRP) may not always reflect ongoing inflammation, especially in patients with non-radiographic axial SpA9. Therefore, accurately measuring the inflammatory burden in Crohn's patients, regardless of musculoskeletal symptoms, is an important area for future research. Initiation of earlier targeted therapy to decrease inflammation may not only prevent incident Crohn's associated SpA, progression of prevalent SpA, with concurrent improvements in HRQoL, but may also improve cardiovascular morbidity and mortality.

In addition, although sacroiliitis is the primary axial feature in SpA, there is increasing evidence that there can also be spinal involvement even in the absence of SI joint inflammation. Recent studies suggest that spinal inflammation can occur in up to one-third of nonradiographic SpA patients with <5 years of disease duration.18 This could be an important early imaging inflammatory biomarker. To our knowledge there are no published studies evaluating spinal and SI joint MRI imaging biomarkers in Crohn's associated SpA.

THE MICROBIOME: A CORRELATE OF INFLAMMATION IN CROHN'S DISEASE? The etiopathogenesis of Crohn's Disease-associated SpA remains a puzzle. As with other autoimmune diseases, interplay between genetic factors such as HLA B27 (Human Leukocyte Antigen- B27) and environmental factors likely play a role. The joint symptoms of SpA are not consistently correlated with bowel disease flares.19 Intestinal microbiota plays a critical role in evolution of our entire immune system, since axenic laboratory animals (germfree animals raised in sterile environment) were noted to have partial restoration of T cell population when these animals are colonized with filamentous bacteria. A symbiotic relationship between the main bacterial phyla is necessary for proper functioning of immune system, since notable alterations in the intestinal microbiome (i.e. dysbiosis) have been suggested in various autoimmune diseases. Reduction in taxa-diversity (such as, enterobacteriaceae, Bacteroidales and Clostridiales) and expansion of certain phyla in the intestine have been recently reported in a large cohort of new onset treatment-naïve Crohn's disease (CD) patients.20 In addition, Dr. Longman's lab has shown that the expansion of immunologically relevant Enterobacteriaceae correlates with Crohn's related SpA among a mixed group of patients with Crohn's and ulcerative colitis, (in press). However, while these are exciting data, SpA cases were identified using a non-validated clinical diagnosis, without systematic rheumatology evaluation and no imaging studies. This will be first study evaluating the microbiome in a carefully phenotyped cohort of Crohn's associated SpA, who will also have detailed MRI imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with biopsy proven Crohn's Disease
2. 50% patients with inflammatory back pain and 50% without inflammatory back pain.
3. Age 18 years and above
4. English Speaking patients only

Exclusion Criteria:

1. History of psoriasis, other inflammatory arthritis
2. No exposure to biologic agent within the past six months (except Vedolizumab, which exerts its effect locally)

2. Contraindication to MRI

3. History of malignancy <5 years in remission, (except for non-melanomatous skin cancer).

4. Non English speaking

5. Unable to comply with study protocol.

6. Critically or terminally ill patients

7. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will biopsy proven Crohn's disease will be enrolled for the study. 50% (15 patients) will have symptoms of inflammatory back pain and 50% will not.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2016-04; Primary Completion 2019-01 (Actual); Study Completion 2021-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Mandl, MD MPH, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lichtenstein GR, Yan S, Bala M, Blank M, Sands BE. Infliximab maintenance treatment reduces hospitalizations, surgeries, and procedures in fistulizing Crohn's disease. Gastroenterology. 2005 Apr;128(4):862-9. doi: 10.1053/j.gastro.2005.01.048. PMID 15825070
- [Background] Bernstein CN, Blanchard JF, Rawsthorne P, Yu N. The prevalence of extraintestinal diseases in inflammatory bowel disease: a population-based study. Am J Gastroenterol. 2001 Apr;96(4):1116-22. doi: 10.1111/j.1572-0241.2001.03756.x. PMID 11316157
- [Background] Dekker-Saeys BJ, Meuwissen SG, Van Den Berg-Loonen EM, De Haas WH, Agenant D, Tytgat GN. Ankylosing spondylitis and inflammatory bowel disease. II. Prevalence of peripheral arthritis, sacroiliitis, and ankylosing spondylitis in patients suffering from inflammatory bowel disease. Ann Rheum Dis. 1978 Feb;37(1):33-5. doi: 10.1136/ard.37.1.33. PMID 629601
- [Background] Shivashankar R, Loftus EV Jr, Tremaine WJ, Bongartz T, Harmsen WS, Zinsmeister AR, Matteson EL. Incidence of spondyloarthropathy in patients with Crohn's disease: a population-based study. J Rheumatol. 2012 Nov;39(11):2148-52. doi: 10.3899/jrheum.120321. Epub 2012 Sep 15. PMID 22984277
- [Background] Bandinelli F, Terenzi R, Giovannini L, Milla M, Genise S, Bagnoli S, Biagini S, Annese V, Matucci-Cerinic M. Occult radiological sacroiliac abnormalities in patients with inflammatory bowel disease who do not present signs or symptoms of axial spondylitis. Clin Exp Rheumatol. 2014 Nov-Dec;32(6):949-52. Epub 2014 Aug 15. PMID 25152017
- [Background] Subramaniam K, Tymms K, Shadbolt B, Pavli P. Spondyloarthropathy in inflammatory bowel disease patients on TNF inhibitors. Intern Med J. 2015 Nov;45(11):1154-60. doi: 10.1111/imj.12891. PMID 26337851
- [Background] Boonen A, Sieper J, van der Heijde D, Dougados M, Bukowski JF, Valluri S, Vlahos B, Kotak S. The burden of non-radiographic axial spondyloarthritis. Semin Arthritis Rheum. 2015 Apr;44(5):556-562. doi: 10.1016/j.semarthrit.2014.10.009. Epub 2014 Oct 22. PMID 25532945
- [Background] Sieper J, van der Heijde D, Dougados M, Mease PJ, Maksymowych WP, Brown MA, Arora V, Pangan AL. Efficacy and safety of adalimumab in patients with non-radiographic axial spondyloarthritis: results of a randomised placebo-controlled trial (ABILITY-1). Ann Rheum Dis. 2013 Jun;72(6):815-22. doi: 10.1136/annrheumdis-2012-201766. Epub 2012 Jul 7. PMID 22772328
- [Background] Sieper J, van der Heijde D. Review: Nonradiographic axial spondyloarthritis: new definition of an old disease? Arthritis Rheum. 2013 Mar;65(3):543-51. doi: 10.1002/art.37803. No abstract available. PMID 23233285
- [Background] Sieper J, Rudwaleit M, Baraliakos X, Brandt J, Braun J, Burgos-Vargas R, Dougados M, Hermann KG, Landewe R, Maksymowych W, van der Heijde D. The Assessment of SpondyloArthritis international Society (ASAS) handbook: a guide to assess spondyloarthritis. Ann Rheum Dis. 2009 Jun;68 Suppl 2:ii1-44. doi: 10.1136/ard.2008.104018. PMID 19433414
- [Background] Sieper J, van der Heijde D, Landewe R, Brandt J, Burgos-Vagas R, Collantes-Estevez E, Dijkmans B, Dougados M, Khan MA, Leirisalo-Repo M, van der Linden S, Maksymowych WP, Mielants H, Olivieri I, Rudwaleit M. New criteria for inflammatory back pain in patients with chronic back pain: a real patient exercise by experts from the Assessment of SpondyloArthritis international Society (ASAS). Ann Rheum Dis. 2009 Jun;68(6):784-8. doi: 10.1136/ard.2008.101501. Epub 2009 Jan 15. PMID 19147614
- [Background] Steer S, Jones H, Hibbert J, Kondeatis E, Vaughan R, Sanderson J, Gibson T. Low back pain, sacroiliitis, and the relationship with HLA-B27 in Crohn's disease. J Rheumatol. 2003 Mar;30(3):518-22. PMID 12610811
- [Background] van Steenbergen HW, Huizinga TW, van der Helm-van Mil AH. The preclinical phase of rheumatoid arthritis: what is acknowledged and what needs to be assessed? Arthritis Rheum. 2013 Sep;65(9):2219-32. doi: 10.1002/art.38013. No abstract available. PMID 23686440
- [Background] Solomon DH, Reed GW, Kremer JM, Curtis JR, Farkouh ME, Harrold LR, Hochberg MC, Tsao P, Greenberg JD. Disease activity in rheumatoid arthritis and the risk of cardiovascular events. Arthritis Rheumatol. 2015 Jun;67(6):1449-55. doi: 10.1002/art.39098. PMID 25776112
- [Background] Roubille C, Richer V, Starnino T, McCourt C, McFarlane A, Fleming P, Siu S, Kraft J, Lynde C, Pope J, Gulliver W, Keeling S, Dutz J, Bessette L, Bissonnette R, Haraoui B. The effects of tumour necrosis factor inhibitors, methotrexate, non-steroidal anti-inflammatory drugs and corticosteroids on cardiovascular events in rheumatoid arthritis, psoriasis and psoriatic arthritis: a systematic review and meta-analysis. Ann Rheum Dis. 2015 Mar;74(3):480-9. doi: 10.1136/annrheumdis-2014-206624. Epub 2015 Jan 5. PMID 25561362
- [Background] Exarchou S, Lie E, Lindstrom U, Askling J, Forsblad-d'Elia H, Turesson C, Kristensen LE, Jacobsson LT. Mortality in ankylosing spondylitis: results from a nationwide population-based study. Ann Rheum Dis. 2016 Aug;75(8):1466-72. doi: 10.1136/annrheumdis-2015-207688. Epub 2015 Sep 2. PMID 26338036
- [Background] Haroon NN, Paterson JM, Li P, Inman RD, Haroon N. Patients With Ankylosing Spondylitis Have Increased Cardiovascular and Cerebrovascular Mortality: A Population-Based Study. Ann Intern Med. 2015 Sep 15;163(6):409-16. doi: 10.7326/M14-2470. PMID 26258401
- [Background] van der Heijde D, Sieper J, Maksymowych WP, Brown MA, Lambert RG, Rathmann SS, Pangan AL. Spinal inflammation in the absence of sacroiliac joint inflammation on magnetic resonance imaging in patients with active nonradiographic axial spondyloarthritis. Arthritis Rheumatol. 2014 Mar;66(3):667-73. doi: 10.1002/art.38283. PMID 24574227
- [Background] Manasson J, Scher JU. Spondyloarthritis and the microbiome: new insights from an ancient hypothesis. Curr Rheumatol Rep. 2015 Feb;17(2):10. doi: 10.1007/s11926-014-0487-7. PMID 25663180
- [Background] Gevers D, Kugathasan S, Denson LA, Vazquez-Baeza Y, Van Treuren W, Ren B, Schwager E, Knights D, Song SJ, Yassour M, Morgan XC, Kostic AD, Luo C, Gonzalez A, McDonald D, Haberman Y, Walters T, Baker S, Rosh J, Stephens M, Heyman M, Markowitz J, Baldassano R, Griffiths A, Sylvester F, Mack D, Kim S, Crandall W, Hyams J, Huttenhower C, Knight R, Xavier RJ. The treatment-naive microbiome in new-onset Crohn's disease. Cell Host Microbe. 2014 Mar 12;15(3):382-392. doi: 10.1016/j.chom.2014.02.005. PMID 24629344

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were identified by physicians in the study at outpatient IBD clinics at Cornell during scheduled visits and through review of medical records. Gastroenterologists at the IBD clinic and HSS rheumatologists were contacted and asked about potential patients. Flyers were placed in patient rooms so patients could express interest in study. We approached potential subjects via postal and/or email addresses and sent survey questionnaire to determine eligibility. Recruitment done 4/2016-5/2017.
Groups:
- Adult Subjects With Crohn's Disease: These were consecutive subjects prospectively identified and enrolled from an outpatient clinic of Jill Roberts Center for Inflammatory Bowel Disease (IBD) at a tertiary care academic medical center. Subjects between 18 and 65 were enrolled from April 2016 through May 2017. All subjects met clinical, pathological or radiological criteria for CD. Patients with ulcerative colitis, indeterminate colitis, other inflammatory arthritis (eg, rheumatoid arthritis, systemic lupus erythematosus, psoriatic or reactive arthritis), co-existent autoimmune diseases (eg, celiac disease, Behçet's disease) or skin psoriasis were excluded. All subjects were either biologic naïve or had been off systemic biologics >6 months prior to enrollment and could remain on non-biologic CD therapy (eg, methotrexate, sulfasalazine, azathioprine or 6-mercaptopurine). Patients could also be on vedolizumab, an antagonist of α4β7 integrin in the intestinal epithelium which has no established efficacy in extra-intestinal manifestations of CD. Other exclusions included malignancy less than 5 years in remission (except for non-melanomatous skin cancer) or having a contraindication to MRI.
Period: Overall Study
Arm/Group | Adult Subjects With Crohn's Disease
Started | 33
Any Back Pain | 19
No Back Pain | 14
MRI Showing Presence of Sacroiliitis | 4
MRI Not Showing Sacroiliitis | 29
Classified as Having Inflammatory Back Pain by the ASAS Criteria | 6
Not Classified as Having Inflammatory Back Pain by the ASAS Criteria | 25
Having Bone Marrow Edema Seen in MRI | 33
Having Erosion (a Structural Lesion) Seen in MRI | 33
Having Fat Metaplasia Seen in MRI | 33
Having Backfill (Type of Structural Lesion) Seen in MRI | 33
Having Ankylosis Seen in MRI | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adult Subjects With Crohn's Disease
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36.4 [27.2 to 49.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 25
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With MRI Positivity- Global Assessment Positive
Description: MRIs were independently read and scored by 2 expert rheumatologists and 1 newly trained rheumatologist reader, blinded to any clinical information. MRIs were evaluated and scored for presence of bone marrow edema (BME) and structural lesions (erosion, fat metaplasia, backfill and ankylosis) using a validated scoring method originally derived from the Spondyloarthritis Research Consortium of Canada SIJ module. MRI was considered "positive" for presence of sacroiliitis if it met global evaluation, based on the reader's overall evaluation of presence or absence of sacroiliitis by taking into account the contextual signature of both active and structural SIJ lesions. For analysis, MRI positivity for sacroiliitis was defined based on majority-of-readers agreement (≥2 out of 3).
Time Frame: one study visit
Measure: Count of Participants; unit: Participants
Groups:
- Any Back Pain: Subjects with Crohn's Disease with back pain.
- No Back Pain: Subjects with Crohn's disease without back pain.
Arm/Group | Any Back Pain | No Back Pain
Number analyzed (Participants) | 19 | 14
Participants | 4 | 0

2. Primary Outcome: Number of Participants With MRI Positivity- ASAS Positive
Description: Assessment of SpondyloArthritis international Society. Subjects are positive if they fulfill 4 out of following 5 back pain parameters: onset of symptoms <40 years of age, insidious onset of pain, nocturnal pain, improvement with exercise and no improvement with rest.
Time Frame: one study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Any Back Pain | No Back Pain
Number analyzed (Participants) | 19 | 14
Participants | 4 | 2

3. Primary Outcome: Number of Participants With MRI Positivity- SPACE Positive
Description: SpondyloArthritis Caught Early. Positivity based on presence of erosions and fat metaplasia.
Time Frame: one study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Any Back Pain | No Back Pain
Number analyzed (Participants) | 19 | 14
Participants | 0 | 0

4. Primary Outcome: Number of Participants With MRI Positivity- Morpho Positive
Description: Positivity based on presence of bone marrow edema (BME) and/or erosion.
Time Frame: one study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Any Back Pain | No Back Pain
Number analyzed (Participants) | 19 | 14
Participants | 5 | 1

5. Secondary Outcome: Number of Participants With Axial Spondyloarthritis Based on European Spondyloarthropathy Study Group (ESSG) Guidelines
Description: Assessment of SpondyloArthritis international Society criteria was utilized to define inflammatory back pain.
Time Frame: one study visit
Population: There is not another Arm with "No Back Pain" because this analysis was not done on any patients who identified as having no back pain, since back pain is the primary symptom of axial spondyloarthritis.
Measure: Count of Participants; unit: Participants
Arm/Group | Any Back Pain
Number analyzed (Participants) | 19
Participants | 13

6. Secondary Outcome: Number of Participants With Current Peripheral Arthritis
Time Frame: one study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Any Back Pain | No Back Pain
Number analyzed (Participants) | 19 | 14
Participants | 14 | 4

7. Secondary Outcome: Number of Participants With a History of Peripheral Arthritis
Time Frame: one study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Any Back Pain | No Back Pain
Number analyzed (Participants) | 19 | 14
Participants | 16 | 6

8. Secondary Outcome: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: Minimum 0. Maximum 10. A score of 0 = none (no symptoms), and a score of 10 = very severe symptoms.
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Any Back Pain | No Back Pain
Number analyzed (Participants) | 19 | 14
score on a scale | 5.3 (1.8) | 2.4 (1.6)

9. Secondary Outcome: Bath Ankylosing Spondylitis Metrology Index (BASMI)
Description: The scale of the BASMI ranges from 0 to 10, where 0 is no mobility limitation and 10 is a very severe limitation.
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Any Back Pain | No Back Pain
Number analyzed (Participants) | 19 | 14
score on a scale | 2.9 (0.9) | 2.1 (0.9)

10. Secondary Outcome: Ankylosing Spondylitis Disease Activity Index C-reactive Protein (ASDAS-CRP)
Description: Ankylosing Spondylitis Disease Activity Index C-reactive protein. Higher score indicates worse symptoms. ASDAS-CRP = 0.12 x Back Pain + 0.06 x Duration of Morning Stiffness + 0.11 x Patient Global + 0.07 x Peripheral Pain/Swelling + 0.58 x Ln(CRP+1)
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Any Back Pain | No Back Pain
Number analyzed (Participants) | 19 | 14
score on a scale | 3.1 (0.9) | 2.1 (0.9)

11. Secondary Outcome: CRP (C-reactive Protein)
Description: Peripheral blood was collected for measurement of CRP.
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Any Back Pain | No Back Pain
Number analyzed (Participants) | 19 | 14
mg/L | 1.6 (2.0) | 1.7 (3.3)

12. Secondary Outcome: Duration of Crohn's Disease for Participants
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Any Back Pain | No Back Pain
Number analyzed (Participants) | 19 | 14
years | 11.9 (6.7) | 14.2 (10.5)

13. Secondary Outcome: Number of Participants Using Vedolizumab for Crohn's Disease
Time Frame: one study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Any Back Pain | No Back Pain
Number analyzed (Participants) | 19 | 13
Participants | 3 | 4

14. Secondary Outcome: Number of Participants With a Past History of Biologic Use for Crohn's Disease
Time Frame: one study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Any Back Pain | No Back Pain
Number analyzed (Participants) | 19 | 13
Participants | 3 | 4

15. Secondary Outcome: Number of Participants Who Have Had Surgery Related to Crohn's Disease
Time Frame: one study visit
Population: The number of participants here only adds up to 31, instead of 33, because data was not collected or lost for two participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Any Back Pain | No Back Pain
Number analyzed (Participants) | 18 | 13
Participants | 10 | 9

16. Secondary Outcome: Crohn's Disease Activity (Harvey Bradshaw Index (HBI) Score)
Description: HBI consists of five parameters, which are all clinical. These parameters are: patient well-being (previous day). abdominal pain (previous day), number of liquid or soft stools (previous day), abdominal mass, and complications.
  Patient well-being is scored with: 0 = very well, 1 = slightly below par, 2 = poor, 3 = very poor, 4 = terrible.
  Abdominal pain is scored as: 0 = none, 1 = mild, 2 = moderate, 3 = severe. Abdominal mass is scored as: 0 = none, 1 = dubious, 2 = definite, 3 = definite and tender.
  Complications can be answered with "No" (0 points) or by choosing from a list, with each selection being 1 point. The list is: arthralgia, uveitis, erythema nodosum, aphthous ulcer, pyoderma gangrenosum, anal fissures, appearance of a new fistula, abscess.
  Calculation formula: sum of the scores of all 5 parameters. < 5 remission 5 - 7 mild activity 8 - 16 moderate activity > 16 severe activity
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Any Back Pain | No Back Pain
Number analyzed (Participants) | 19 | 14
score on a scale | 9.1 (4.9) | 6.9 (3.7)

17. Secondary Outcome: Number of Participants With Inflammatory Back Pain
Time Frame: one study visit
Measure: Count of Participants; unit: Participants
Groups:
- Global MRI Positive: MRI showed evidence of sacroiliitis.
- Global MRI Negative: MRI did not show evidence of sacroiliitis.
Arm/Group | Global MRI Positive | Global MRI Negative
Number analyzed (Participants) | 4 | 29
Participants | 4 | 15

18. Secondary Outcome: Number of Participants With Current Peripheral Arthritis
Time Frame: one study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Global MRI Positive | Global MRI Negative
Number analyzed (Participants) | 4 | 29
Participants | 3 | 15

19. Secondary Outcome: Number of Participants With a History of Peripheral Arthritis
Time Frame: one study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Global MRI Positive | Global MRI Negative
Number analyzed (Participants) | 4 | 29
Participants | 4 | 18

20. Secondary Outcome: Number of Participants With Current Enthesitis
Time Frame: one study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Global MRI Positive | Global MRI Negative
Number analyzed (Participants) | 4 | 29
Participants | 1 | 8

21. Secondary Outcome: Number of Participants With a History of Uveitis
Time Frame: one study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Global MRI Positive | Global MRI Negative
Number analyzed (Participants) | 4 | 29
Participants | 1 | 3

22. Secondary Outcome: Number of Participants With a History of Dactylitis
Time Frame: one study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Global MRI Positive | Global MRI Negative
Number analyzed (Participants) | 4 | 29
Participants | 2 | 1

23. Secondary Outcome: Number of Participants With HLA-B27 (Human Leukocyte Antigen B-27)
Time Frame: one study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Global MRI Positive | Global MRI Negative
Number analyzed (Participants) | 4 | 29
Participants | 0 | 1

24. Secondary Outcome: CRP (C-reactive Protein)
Description: Peripheral blood was collected for measurement of CRP.
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Global MRI Positive | Global MRI Negative
Number analyzed (Participants) | 4 | 29
mg/L | 2.6 (3.0) | 1.5 (2.6)

25. Secondary Outcome: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: Minimum 0. Maximum 10. A score of 0 = none (no symptoms), and a score of 10 = very severe symptoms.
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Global MRI Positive | Global MRI Negative
Number analyzed (Participants) | 4 | 29
score on a scale | 4.3 (1.7) | 4.2 (2.4)

26. Secondary Outcome: Bath Ankylosing Spondylitis Metrology Index (BASMI)
Description: The scale of the BASMI ranges from 0 to 10, where 0 is no mobility limitation and 10 is a very severe limitation.
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Global MRI Positive | Global MRI Negative
Number analyzed (Participants) | 4 | 29
score on a scale | 4.1 (0.7) | 2.4 (0.8)

27. Secondary Outcome: Ankylosing Spondylitis Disease Activity Index C-reactive Protein (ASDAS-CRP)
Description: A higher score indicates worse symptoms. ASDAS-CRP = 0.12 x Back Pain + 0.06 x Duration of Morning Stiffness + 0.11 x Patient Global + 0.07 x Peripheral Pain/Swelling + 0.58 x Ln(CRP+1)
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Global MRI Positive | Global MRI Negative
Number analyzed (Participants) | 4 | 29
score on a scale | 3.3 (0.4) | 2.5 (1.2)

28. Secondary Outcome: Duration of Crohn's Disease
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Global MRI Positive | Global MRI Negative
Number analyzed (Participants) | 4 | 29
years | 17.9 (3.8) | 12.2 (8.7)

29. Secondary Outcome: Crohn's Disease Activity (Harvey Bradshaw Index (HBI) Score)
Description: as for outcome 16
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Global MRI Positive | Global MRI Negative
Number analyzed (Participants) | 4 | 29
score on a scale | 7.8 (4.9) | 8.3 (4.5)

30. Secondary Outcome: Number of Participants Using Vedolizumab for Crohn's Disease
Time Frame: one study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Global MRI Positive | Global MRI Negative
Number analyzed (Participants) | 4 | 28
Participants | 0 | 7

31. Secondary Outcome: Number of Participants With a Prior History of Biologic Use for Crohn's Disease
Time Frame: one study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Global MRI Positive | Global MRI Negative
Number analyzed (Participants) | 4 | 28
Participants | 3 | 16

32. Secondary Outcome: Number of Participants Who Have Had Surgery Related to Crohn's Disease
Time Frame: one study visit
Measure: Count of Participants; unit: Participants
Arm/Group | Global MRI Positive | Global MRI Negative
Number analyzed (Participants) | 4 | 28
Participants | 3 | 16

33. Secondary Outcome: Interleukin 2
Description: Concentration of IL-2 in peripheral blood of participants.
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- ASAS (Assessment of SpondyloArthritis International Society) MRI Positive: Subjects classified as having inflammatory back pain for meeting 4 out of the 5 following back pain parameters: onset of symptoms <40 years of age, insidious onset of pain, nocturnal pain, improvement with exercise and no improvement with rest.
- ASAS (Assessment of SpondyloArthritis International Society) MRI Negative: Subjects not classified as having inflammatory back pain for meeting 4 out of the 5 following back pain parameters: onset of symptoms <40 years of age, insidious onset of pain, nocturnal pain, improvement with exercise and no improvement with rest.
Arm/Group | ASAS (Assessment of SpondyloArthritis International Society) MRI Positive | ASAS (Assessment of SpondyloArthritis International Society) MRI Negative
Number analyzed (Participants) | 6 | 25
pg/mL | 4.7 (2.0) | 5.6 (7.8)

34. Secondary Outcome: Interleukin 4
Description: Concentration of IL-4 in peripheral blood of participants.
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | ASAS (Assessment of SpondyloArthritis International Society) MRI Positive | ASAS (Assessment of SpondyloArthritis International Society) MRI Negative
Number analyzed (Participants) | 6 | 25
pg/mL | 3.5 (1.6) | 5.7 (4.6)

35. Secondary Outcome: Interleukin 5
Description: Concentration of IL-5 in peripheral blood of participants.
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | ASAS (Assessment of SpondyloArthritis International Society) MRI Positive | ASAS (Assessment of SpondyloArthritis International Society) MRI Negative
Number analyzed (Participants) | 6 | 25
pg/mL | 3.7 (0.0) | 3.8 (0.1)

36. Secondary Outcome: Interleukin 6
Description: Concentration of IL-6 in peripheral blood of participants.
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | ASAS (Assessment of SpondyloArthritis International Society) MRI Positive | ASAS (Assessment of SpondyloArthritis International Society) MRI Negative
Number analyzed (Participants) | 6 | 25
pg/mL | 6.2 (7.2) | 5.1 (6.9)

37. Secondary Outcome: Interleukin 9
Description: Concentration of IL-9 in peripheral blood of participants.
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | ASAS (Assessment of SpondyloArthritis International Society) MRI Positive | ASAS (Assessment of SpondyloArthritis International Society) MRI Negative
Number analyzed (Participants) | 6 | 25
pg/mL | 2.4 (1.5) | 1.9 (0.9)

38. Secondary Outcome: Interleukin 10
Description: Concentration of IL-10 in peripheral blood of participants.
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | ASAS (Assessment of SpondyloArthritis International Society) MRI Positive | ASAS (Assessment of SpondyloArthritis International Society) MRI Negative
Number analyzed (Participants) | 6 | 25
pg/mL | 31.0 (59.3) | 6.5 (1.8)

39. Secondary Outcome: Interleukin 13
Description: Concentration of IL-13 in peripheral blood of participants.
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | ASAS (Assessment of SpondyloArthritis International Society) MRI Positive | ASAS (Assessment of SpondyloArthritis International Society) MRI Negative
Number analyzed (Participants) | 6 | 25
pg/mL | 8.9 (6.3) | 8.9 (4.4)

40. Secondary Outcome: Interleukin 12-23
Description: Concentration of IL 12-23 in peripheral blood of participants.
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | ASAS (Assessment of SpondyloArthritis International Society) MRI Positive | ASAS (Assessment of SpondyloArthritis International Society) MRI Negative
Number analyzed (Participants) | 6 | 25
pg/mL | 214.0 (159.5) | 259.1 (227.7)

41. Secondary Outcome: Interleukin 17A
Description: Concentration of IL-17A in peripheral blood of participants.
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | ASAS (Assessment of SpondyloArthritis International Society) MRI Positive | ASAS (Assessment of SpondyloArthritis International Society) MRI Negative
Number analyzed (Participants) | 6 | 25
pg/mL | 25.3 (13.1) | 21.1 (10.5)

42. Secondary Outcome: Interleukin 17F
Description: Concentration of IL-17F in peripheral blood of participants.
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | ASAS (Assessment of SpondyloArthritis International Society) MRI Positive | ASAS (Assessment of SpondyloArthritis International Society) MRI Negative
Number analyzed (Participants) | 6 | 25
pg/mL | 4.8 (2.2) | 3.8 (3.5)

43. Secondary Outcome: Interleukin 21
Description: Concentration of IL-21 in peripheral blood of participants.
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | ASAS (Assessment of SpondyloArthritis International Society) MRI Positive | ASAS (Assessment of SpondyloArthritis International Society) MRI Negative
Number analyzed (Participants) | 6 | 25
pg/mL | 19.8 (36.2) | 40.0 (43.2)

44. Secondary Outcome: Interleukin 22
Description: Concentration of IL-22 in peripheral blood of participants.
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | ASAS (Assessment of SpondyloArthritis International Society) MRI Positive | ASAS (Assessment of SpondyloArthritis International Society) MRI Negative
Number analyzed (Participants) | 6 | 25
pg/mL | 15.2 (7.1) | 16.7 (11.2)

45. Secondary Outcome: Interferon-γ
Description: Concentration of INFγ in peripheral blood of participants.
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | ASAS (Assessment of SpondyloArthritis International Society) MRI Positive | ASAS (Assessment of SpondyloArthritis International Society) MRI Negative
Number analyzed (Participants) | 6 | 25
pg/mL | 75.7 (31.0) | 79.0 (28.8)

46. Secondary Outcome: TNF-α (Tumor Necrosis Factor)
Description: Concentration of TNF-α in peripheral blood of participants.
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | ASAS (Assessment of SpondyloArthritis International Society) MRI Positive | ASAS (Assessment of SpondyloArthritis International Society) MRI Negative
Number analyzed (Participants) | 6 | 25
pg/mL | 19.5 (15.2) | 35.4 (94.1)

47. Secondary Outcome: Mean Number of Sacroiliac Joint (SIJ) Quadrants Affected by BME or Structural Lesions for Each Participant
Description: MRIs were independently read and scored by 2 expert rheumatologists and 1 newly trained rheumatologist reader, blinded to any clinical information. MRIs were evaluated and scored for presence of bone marrow edema (BME) and structural lesions (erosion, fat metaplasia, backfill and ankylosis) using a validated scoring method originally derived from the Spondyloarthritis Research Consortium of Canada SIJ module. Readers determined whether BME and the structural lesions were present in each of the quadrants for each participant. There are 2 sacroiliac joints and 4 quadrants for each joint, for a total of 8 quadrants for each participant.
Time Frame: one study visit
Measure: Mean (Standard Deviation); unit: Number of Quadrants Affected per Person
Groups:
- Bone Marrow Edema: Type of lesion seen in MRI.
- Erosion; Fat Metaplasia; Backfill; Ankylosis: Type of structural lesion seen in MRI.
Arm/Group | Bone Marrow Edema | Erosion | Fat Metaplasia | Backfill | Ankylosis
Number analyzed (Participants) | 33 | 33 | 33 | 33 | 33
Number of Quadrants Affected per Person | 0.86 (1.45) | 0.05 (0.15) | 0.98 (3.55) | 0.04 (0.23) | 1.02 (3.45)

48. Secondary Outcome: Median Number of Sacroiliac Joint (SIJ) Quadrants Affected by BME or Structural Lesions for Each Participant
Description: as for outcome 47
Time Frame: one study visit
Measure: Median (Inter-Quartile Range); unit: Number of Quadrants Affected per Person
Arm/Group | Bone Marrow Edema | Erosion | Fat Metaplasia | Backfill | Ankylosis
Number analyzed (Participants) | 33 | 33 | 33 | 33 | 33
Number of Quadrants Affected per Person | 0 [0 to 1.3] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

49. Secondary Outcome: Number of Participants With ≥1 Quadrant Affected by BME or Structural Lesions
Description: MRIs were independently read and scored by 2 expert rheumatologists and 1 newly trained rheumatologist reader, blinded to any clinical information. MRIs were evaluated and scored for presence of bone marrow edema (BME) and structural lesions (erosion, fat metaplasia, backfill and ankylosis) using a validated scoring method originally derived from the Spondyloarthritis Research Consortium of Canada SIJ module. Readers determined whether BME and the structural lesions were present in each of the quadrants for each participant. There are 2 sacroiliac joints and 4 quadrants for each joint, for a total of 8 quadrants for each participant. A quadrant is deemed affected if concordantly reported by ≥ 2/3 readers.
Time Frame: one study visit
Population: These Arms/Groups indicate which specific lesion is being looked at in the MRIs by the readers. Each of the 33 participants in the trial had their MRIs looked at for each of the lesions, therefore the overall number of participants analyzed is 33 for each Arm/Group. The count of participants indicates how many participants had at least 1 quadrant affected by a given lesion.
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Edema | Erosion | Fat Metaplasia | Backfill | Ankylosis
Number analyzed (Participants) | 33 | 33 | 33 | 33 | 33
Participants | 10 | 1 | 2 | 1 | 2

50. Secondary Outcome: Number of Participants With ≥2 Quadrants Affected by BME or Structural Lesions
Description: as for outcome 49
Time Frame: one study visit
Population: These Arms/Groups indicate which specific lesion is being looked at in the MRIs by the readers. Each of the 33 participants in the trial had their MRIs looked at for each of the lesions, therefore the overall number of participants analyzed is 33 for each Arm/Group. The count of participants indicates how many participants had at least 2 quadrants affected by a given lesion.
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Edema | Erosion | Fat Metaplasia | Backfill | Ankylosis
Number analyzed (Participants) | 33 | 33 | 33 | 33 | 33
Participants | 7 | 0 | 1 | 0 | 2

51. Secondary Outcome: Number of Participants With ≥3 Quadrants Affected by BME or Structural Lesions
Description: as for outcome 49
Time Frame: one study visit
Population: These Arms/Groups indicate which specific lesion is being looked at in the MRIs by the readers. Each of the 33 participants in the trial had their MRIs looked at for each of the lesions, therefore the overall number of participants analyzed is 33 for each Arm/Group. The count of participants indicates how many participants had at least 3 quadrants affected by a given lesion.
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Edema | Erosion | Fat Metaplasia | Backfill | Ankylosis
Number analyzed (Participants) | 33 | 33 | 33 | 33 | 33
Participants | 5 | 0 | 1 | 0 | 2

52. Secondary Outcome: Number of Participants With ≥4 Quadrants Affected by BME or Structural Lesions
Description: as for outcome 49
Time Frame: one study visit
Population: These Arms/Groups indicate which specific lesion is being looked at in the MRIs by the readers. Each of the 33 participants in the trial had their MRIs looked at for each of the lesions, therefore the overall number of participants analyzed is 33 for each Arm/Group. The count of participants indicates how many participants had at least 4 quadrants affected by a given lesion.
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Edema | Erosion | Fat Metaplasia | Backfill | Ankylosis
Number analyzed (Participants) | 33 | 33 | 33 | 33 | 33
Participants | 2 | 0 | 1 | 0 | 2

53. Secondary Outcome: Number of Participants With ≥6 Quadrants Affected by BME or Structural Lesions
Description: as for outcome 49
Time Frame: one study visit
Population: These Arms/Groups indicate which specific lesion is being looked at in the MRIs by the readers. Each of the 33 participants in the trial had their MRIs looked at for each of the lesions, therefore the overall number of participants analyzed is 33 for each Arm/Group. The count of participants indicates how many participants had at least 6 quadrants affected by a given lesion.
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Edema | Erosion | Fat Metaplasia | Backfill | Ankylosis
Number analyzed (Participants) | 33 | 33 | 33 | 33 | 33
Participants | 1 | 0 | 1 | 0 | 2

54. Secondary Outcome: Number of Participants With ≥5 Quadrants Affected by BME or Structural Lesions
Description: as for outcome 49
Time Frame: one study visit
Population: These Arms/Groups indicate which specific lesion is being looked at in the MRIs by the readers. Each of the 33 participants in the trial had their MRIs looked at for each of the lesions, therefore the overall number of participants analyzed is 33 for each Arm/Group. The count of participants indicates how many participants had at least 5 quadrants affected by a given lesion.
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Edema | Erosion | Fat Metaplasia | Backfill | Ankylosis
Number analyzed (Participants) | 33 | 33 | 33 | 33 | 33
Participants | 2 | 0 | 1 | 0 | 2

55. Secondary Outcome: Number of Participants With ≥7 Quadrants Affected by BME or Structural Lesions
Description: as for outcome 49
Time Frame: one study visit
Population: These Arms/Groups indicate which specific lesion is being looked at in the MRIs by the readers. Each of the 33 participants in the trial had their MRIs looked at for each of the lesions, therefore the overall number of participants analyzed is 33 for each Arm/Group. The count of participants indicates how many participants had at least 7 quadrants affected by a given lesion.
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Edema | Erosion | Fat Metaplasia | Backfill | Ankylosis
Number analyzed (Participants) | 33 | 33 | 33 | 33 | 33
Participants | 0 | 0 | 1 | 0 | 2

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Adult Subjects With Crohn's Disease
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT02709694/Prot_SAP_000.pdf
  • Informed Consent Form (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT02709694/ICF_001.pdf